CLINICAL TRIAL: NCT00642824
Title: Local Substudy Associated to the International Study MO19390 to Determine the BRCA1 Gene mRNA Expression as a Predictive Marker of Response to Chemotherapy
Brief Title: A Genetic Substudy Associated With the Avastin (Bevacizumab) Study MO19390 in Patients With Advanced or Recurrent Non-Squamous Cell Lung Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low enrollment. No statistical analyses were performed.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21150
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Standard chemotherapy; Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: Standard chemotherapy — As prescribed--chemotherapy may be a)gemcitabine/cisplatin, b)vinorelbine + cisplatin/docetaxel + cisplatin or c)vinorelbine or docetaxel.
Drug: bevacizumab [Avastin] — 15mg/kg iv or 7.5mg/kg on day 1, and subsequently once every 3 weeks

SUMMARY:
This single arm genetic substudy of MO19390 will test the hypothesis that there is a positive relationship between mRNA BRCAI levels and the response to different chemotherapy combinations plus Avastin. A subset of patients participating in MO19390, and receiving Avastin 15mg/kg iv on day 1 and subsequently once every 3 weeks, will undergo BRCAI mRNA expression determination. Depending on the BRCAI mRNA level (low, medium or high) they will receive a different chemotherapy regimen in combination with Avastin: a)gemcitabine/cisplatin, b)vinorelbine + cisplatin/docetaxel + cisplatin or c)vinorelbine or docetaxel. Avastin treatment will continue after completion of chemotherapy cycles until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* participating in, and meeting all inclusion/exclusion criteria of, MO19390.

Exclusion Criteria:

* not meeting the inclusion/exclusion criteria of MO19390.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Event driven

SECONDARY OUTCOMES:
Overall survival; response rates | Event driven
Adverse events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Spain (19):
  - Alcorcón
  - Alcoy
  - Alicante
  - Badalona
  - Barakaldo
  - Burgos
  - Elche
  - Girona
  - Huesca
  - Las Palmas de Gran Canaria
  - Lugo
  - Madrid
  - Murcia
  - Palma de Mallorca
  - Pamplona
  - Salamanca
  - San Cristóbal de La Laguna
  - Valencia
  - Zaragoza